

# Statistical Analysis Plan

Protocol No.: JS-OAP2-US01, Version 6.0

A Phase 2, Double-Blind, Randomized, Controlled Study to Evaluate the Efficacy and Safety of JointStem, Autologous Adipose Tissue Derived Mesenchymal Stem Cells, in Treatment of Osteoarthritis

Sponsor: Nature Cell Co., Ltd

Protocol Version: JS-OAP2-US01, Version 6.0, April 07, 2017

SAP Version No & Date: SAP\_JS-OAP2-US01, Version 2.0, April 05, 2018

Version: 2.0 



# **Signature Page**

| Prepared by: | |
|------------------------------------------|-------------------|
| Ami Yu STAT Manager, HERINGS | Date (DD/MM/YYYY) |
| Reviewed by: | |
| Byung-Ho Nam STAT Director, HERINGS | Date (DD/MM/YYYY) |
| Hugh Lee Project Director, KCRN Research | Date (DD/MM/YYYY) |
| Approval by: | |
| Title, Signature<br>Sponsor | Date (DD/MM/YYYY) |



# TABLE OF CONTENTS

| AB | BREV | IATIONS | 5 |
|---|---|---|---|
| 1. | INT | RODUCTION | 6 |
| | 1.1 | STUDY OBJECTIVES | 6 |
| | | 1.1.1 Primary Objective | 6 |
| | 1.2 | STUDY ENDPOINTS | 6 |
| | | 1.2.1 Primary Efficacy Endpoints | 6 |
| | | <ul><li>1.2.2 Secondary Efficacy Endpoints</li><li>1.2.3 Safety Endpoints</li></ul> | 6<br>7 |
| | 1.3 | SUMMARY OF THE STUDY DESIGN | 7 |
| | -10 | 1.3.1 General Study Design and Plan | 7 |
| | | 1.3.2 Randomization and Blinding | 9 |
| | | 1.3.3 Sample Size and Statistical Power Considerations | 9 |
| 2 | OT A | 1.3.4 Interim Analysis | 9 |
| 2. | SIA | TISTICAL METHODS | 9 |
| | 2.1 | GENERAL CONSIDERATIONS | 9 |
| | 2.2 | 2.1.1 Reporting Precision | 10 |
| | 2.2 | DEFINITIONS OF ANALYSIS POPULATIONS (ANALYSIS SETS) 2.2.1 Intention-To-Treat Population (ITT) | 10<br>10 |
| | | 2.2.2 Per-Protocol Population (PP) | 10 |
| | | 2.2.3 Safety Population | 10 |
| | 2.3 | TIME WINDOWS FOR ANALYSIS | 10 |
| | 2.4 | HANDLING OF MISSING DATA | 11 |
| | 2.5 | Analysis software | 11 |
| 3. | STU | DY SUBJECTS | 11 |
| | 3.1 | DISPOSITION OF SUBJECTS | 11 |
| | 3.2 | PROTOCOL DEVIATIONS | 11 |
| 4. | DEM | MOGRAPHICS AND BASELINE CHARACTERISTICS | 11 |
| | 4.1 | DEMOGRAPHICS AND BASELINE CHARACTERISTICS | 11 |
| | 4.2 | MEDICAL HISTORY | 12 |
| 5. | STU | DY DRUG AND EXPOSURE | 12 |
| | 5.1 | Treatment | 12 |
| | 5.2 | PRIOR AND CONCOMITANT THERAPY | 12 |
| 6. | EFF. | ICACY ANALYSES | 12 |
| | 6.1 | PRIMARY EFFICACY ANALYSIS | 13 |
| | 6.2 | SECONDARY EFFICACY ANALYSIS | 14 |
| | | 6.2.1 WOMAC Score | 14 |
| | | 6.2.2 VAS Score | 15 |

Sponsor: Nature Cell Co., Ltd **HERINGS** Statistical Analysis Plan V2.0 6.2.3 MRI 15 6.2.4 Lysholm Knee Scoring Scale 16 6.2.5 KOOS 16 6.2.6 IKDC 17 6.2.7 RAND-36 Score 17 SAFETY ANALYSIS 7. 18 7.1 ADVERSE EVENTS 18 7.1.1 Deaths, Serious and Other Significant Adverse Events 19 CLINICAL LABORATORY PARAMETERS 7.2 20 7.3 VITAL SIGNS, PHYSICAL EXAMINATIONS FINDINGS, ECG 20 7.3.1 Vital Signs 20 **Physical Examinations** 7.3.2 20 7.3.3 ECG 21 INTERIM ANALYSES AND DATA AND SAFETY MONITORING BOARD 8. (DSMB) 21 8.1 21 **INTERIM ANALYSES** 8.2 **DSMB** 21 9. SUMMARY OF MAJOR CHANGES IN THE PLANNED ANALYSES 21



# **ABBREVIATIONS**

| Abbreviation | Term |
|--------------|-----------------------------------------------------------|
| AdMSC | Adipose Tissue Derived Mesenchymal Stem Cell |
| AEs | Adverse Events |
| ALT | Alanine Aminotransferase |
| ANCOVA | Analysis of Covariance |
| AST | Aspartate Aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| BMI | Body Mass Index |
| BP | Blood Pressure |
| BUN | Blood Urea Nitrogen |
| DSMB | Data and Safety Monitoring Board |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| IKDC | International Knee Documentation Committee |
| ITT | Intention-to-Treat |
| KOOS | Knee Injury & Osteoarthritis Outcome Score |
| LS Means | Least square adjusted means |
| LOCF | Last-Observation-Carry-Forward |
| MedDRA | Medical Dictionary For Regulatory Activities |
| MRI | Magnetic Resonance Imaging |
| PP | Per Protocol |
| PT | Preferred Term |
| PT-INR | Prothrombin Time - International Normalized Ratio |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SI | Système International |
| SOC | System Organ Class |
| TEAE | Treatment-Emergent Adverse Event |
| VAS | Visual Analog Scale |
| WHO | World Health Organization |
| WOMAC | Western Ontario and McMaster Universities Arthritis Index |



#### 1. INTRODUCTION

The purpose of this statistical analysis plan (SAP) is to describe the procedures and the statistical methods that will be used to analyze and report results for Protocol JS-OAP2-US01. This SAP has been developed based on the study protocol (Version 5.0 dated on February 10, 2017) and electronic case report forms (eCRFs) and has been updated according to the amendment of study protocol (Version 6.0, June 26, 2017).

#### 1.1 STUDY OBJECTIVES

# 1.1.1 Primary Objective

The primary objective of the study is to evaluate the efficacy and safety of autologous adipose tissue derived mesenchymal stem cells (AdMSC) for the treatment of osteoarthritis.

#### 1.2 STUDY ENDPOINTS

# 1.2.1 Primary Efficacy Endpoints

The co-primary endpoints are:

Using the following three co-primary efficacy variables, the joint functional improvement of knee joint will be evaluated and gatekeeping procedures will be used for these three hypothesis tests.

- 1) Change of WOMAC score from baseline at Month 6 (JointStem group)
- 2) Change of VAS score from baseline at Month 6 (JointStem group)
- 3) MRI improvement evaluation at Month 6 (JointStem group)

MRI improvement evaluation will be finally analyzed through the following two steps:

- Radiologist will compare and analyze MRI results before and after the administration of IP and write a report for each subject.
- Principal Investigator will evaluate MRI results of subjects as one of three conditions (a: improvement, b: no change, c: progress) based on the radiologist's report stated above.

#### 1.2.2 Secondary Efficacy Endpoints

The secondary efficacy endpoints are:




- 1) JointStem group vs. positive control group
  - ① Change of WOMAC score from baseline at Month 6
  - ② Change of VAS score from baseline at Month 6
  - 3 Change of KOOS from baseline at Month 6
  - Change of Lysholm Knee Scoring Scale from baseline at Month 6
  - © Change of IKDC from baseline at Month 6
  - © Change of RAND-36 Score from baseline at Month 6

# 2) JointStem group

- ① Change of WOMAC score from baseline at Months 9 and 12
- ② Change of VAS score from baseline at Months 9 and 12
- 3 Comparison of MRI improvement evaluations between at Month 6 and at Months 12
- ① Change of Lysholm Knee Scoring Scale from baseline at Months 6, 9 and 12
- © Change of KOOS from baseline at Months 6, 9 and 12
- © Change of IKDC from baseline at Months 6, 9 and 12
- © Change of RAND-36 Score from baseline at Months 6, 9 and 12

# 1.2.3 Safety Endpoints

Safety endpoints include:

- Clinical laboratory tests
- 12-lead Electrocardiogram (ECG)
- Physical examinations
- Vital signs
- Adverse events (AEs) and concomitant medications

#### 1.3 SUMMARY OF THE STUDY DESIGN

#### 1.3.1 General Study Design and Plan

This is a double-blind, randomized, controlled study to evaluate the efficacy and safety of JointStem for the treatment of osteoarthritis. Following a 2-week screening period, approximately 30 subjects will be randomly assigned into one of the following two arms in a 2:1 ratio (2 JointStem: 1 positive control):

- JointStem (1x10<sup>8</sup> cells/3mL)
- Positive control: Hyaluronic Acid

After each subject completes 6-month visit (Visit 6) and the data management team confirms all individual data have no issue, the individual database will be locked and the blinding will be




open for the statistical analysis. Only subjects who are randomized to JointStem group will then be scheduled for 9-month and 12-month follow-up visits (Visits 7 and 8).

The Schedule of Assessments is presented by Table 1.

**Table 1 Schedule of Assessments** 

| | Screen. | Harv. | Treat. | | 1 <sup>st</sup> Fol | low-up | ) | 2 <sup>nd</sup> F | Follow-Up |
|---|---|---|---|---|---|---|---|---|---|
| Blinding | N/A | Double Blinding | | | Open <sup>7</sup> | | | | |
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | ET | 7 | 8 |
| Week / Month | W-7 | W-5 | 0 | M1 | М3 | M6 | <m6< th=""><th>M9</th><th>M12 or<br/>Final FU<sup>6</sup></th></m6<> | M9 | M12 or<br>Final FU <sup>6</sup> |
| Informed consent | X | | | | | | | | |
| Medical and Medication History | X | X | | | | | | | |
| Demographic information | X | | | | | | | | |
| Complete physical examination | X | | X | | X | X | $X^4$ | X | X |
| Vital signs and weight | X | X | X | X | X | X | X | X | X |
| Hematology, serum chemistry, and urinalysis <sup>1</sup> | X | | X | X | X | X | $X^4$ | X | X |
| Pregnancy test <sup>2</sup> | X | | | | | X | $X^4$ | | X |
| HIV test for Screening | X | | | | | | | | |
| 12-lead ECG | X | | X | | | X | $X^4$ | | X |
| X-ray | X | | | | | | | | |
| Eligibility confirmation | X | X | | | | | | | |
| Randomization | | X | | | | | | | |
| Liposuction | | X | | | | | | | |
| Injection of final drug product | | | X | | | | | | |
| AE and concomitant medication assessment | | | X | X | X | X | X | X | X |
| MRI scan <sup>3</sup> | X | | | | | X | $X^5$ | | X |
| WOMAC | | | X | X | X | X | $X^4$ | X | X |
| VAS | X | | X | X | X | X | $X^4$ | X | X |
| Lysholm | | | X | X | X | X | $X^4$ | X | X |
| KOOS | | | X | X | X | X | $X^4$ | X | X |
| IKDC | | | X | X | X | X | $X^4$ | X | X |
| Quality of Life (RAND-36) | | | X | | X | X | $X^4$ | X | X |

- 1. See Appendix 1 for the complete list of laboratory tests
- 2. Serum pregnancy test is performed for all females of childbearing potential (please refer to the relevant inclusion criteria)
- 3. May be performed the day of Visit 2 or after due to scheduling or re-scanning.
- 4. Performed only if the early termination is after V3.
- 5. Performed only if the early termination is after V4.
- 6. Performed if the follow-up is discontinued after V6.
- 7. Only for JointStem group.




# 1.3.2 Randomization and Blinding

As this is a double-blinded study, blinding of the drug contents from the subjects, investigators, and other study personnel at each clinical site is necessary. Because two syringes of JointStem and positive control are different, one physician must be only assigned to the role of syringe injection in order to maintain the double-blinding against other site physicians and staffs.

A subject will be assigned with one randomization code on Visit 2 (Week -5). After each subject completes Visit 6 (Month 6) and the data management team confirms all data have no issue, the randomization codes will be open for the statistical analysis.

A code-break envelope for each subject including the randomization code information will be retained by each site and can be opened, revealing the randomization information, for emergency purposes only. Investigator should note that the occurrence of a serious adverse event (SAE) should not routinely precipitate immediate unblinding. An attempt to contact the sponsor must be made prior to unblinding. If unblinding occurs, the subject must be early terminated; a written explanation must be prepared immediately.

# 1.3.3 Sample Size and Statistical Power Considerations

There was no formal sample size calculation since this is a proof-of-concept study and is not a hypothesis-driven study. The number of enrolled subjects is predefined at n=30, for 20 subjects per study group and 10 subjects per control group.

#### 1.3.4 Interim Analysis

When at least 15 subjects complete 6-month visits (Visit 6, Month 6), one unblinded interim analysis can be performed to evaluate the efficacy and safety of JointStem without the suspension of subject enrollment. No adjustment on the overall alpha-level will be made, as this is not a statistically powered study. The interim analysis is not covered by this SAP.

# 2. STATISTICAL METHODS

#### 2.1 GENERAL CONSIDERATIONS

In general, continuous variables will be summarized by number of subjects, mean, SD, median, minimum, and maximum values. Categorical variables will be summarized by counts and percentage of subjects in each category. Source data for the summary tables and statistical analyses will be presented as subject data listings, which include data collected on the electronic case report forms (eCRFs) as well as any derived variables for all enrolled subjects.




# 2.1.1 Reporting Precision

Summary statistics will be presented to the following degree of precision, unless otherwise specified:

| Statistics | Degree of Precision |
|---|---|
| Mean, Geometric mean, Median, | One decimal place more than the raw data. |
| Quartiles, Confidence limit boundaries | |
| Standard deviation, Standard error | Two decimal places more than the raw data. |
| Minimum, Maximum | The same as the raw data. |
| p-value | Rounded to 4 decimal places and therefore presented |
| | as 0.xxxx; p-values smaller than 0.0001 as '<0.0001'; |
| | p-values greater than 0.9999 as '>0.9999'. |
| Percentage | One decimal place. A percentage of 100% will be |
| | reported as 100%. Percentages of zero will be |
| | reported as 0. |

For weight and height, one decimal place will be used for summary statistics. Fractional numeric values will be presented with a zero to the left of the decimal point (for example, 0.12 - 0.30).

# 2.2 DEFINITIONS OF ANALYSIS POPULATIONS (ANALYSIS SETS)

# 2.2.1 Intention-To-Treat Population (ITT)

An intention-to-treat (ITT) population will include subjects who received the intra-articular injection and have at least post-injection efficacy measurements.

#### 2.2.2 Per-Protocol Population (PP)

All subjects valid for ITT who completed Visit 6 (Month 6) will be 'valid per protocol' (also called 'valid for efficacy'). Additional criteria may be added prior to unblinding the study database.

# 2.2.3 Safety Population

A Safety population will include any subject who was randomized and completed Visit 2 (Week - 5, at which time adipose tissue was be harvested).

# 2.3 TIME WINDOWS FOR ANALYSIS

For by visit safety or efficacy summaries, only scheduled visits will be analyzed.




## 2.4 HANDLING OF MISSING DATA

Last observation carried forward (LOCF) imputation method will be used for efficacy variables, but no adjustments for missing data and no imputation methods are planned for safety variables.

#### 2.5 ANALYSIS SOFTWARE

All summaries and statistical analyses will be generated using SAS® version 9.24 or later.

#### 3. STUDY SUBJECTS

#### 3.1 DISPOSITION OF SUBJECTS

Disposition will be summarized by treatment and total in all enrolled subjects.

The disposition will include the following:

- Subjects Randomized
- Subjects in the ITT Population
- Subjects in the PP Population
- Subjects in the Safety Population
- Subjects completed 6-month follow-up
  - o If No, Reasons for withdrawal
- Subjects completed 12-month follow-up
  - o If No, Reasons for withdrawal

A listing of dispositions will be provided for all enrolled subjects.

# 3.2 PROTOCOL DEVIATIONS

The clinical team will identify deviations and the deviations will be recorded into the database. A subject data listing will be provided.

#### 4. DEMOGRAPHICS AND BASELINE CHARACTERISTICS

#### 4.1 DEMOGRAPHICS AND BASELINE CHARACTERISTICS

Demographic data (age, gender, race, and ethnicity) and baseline characteristics (including height, weight and body mass index (BMI)) collected at study screening will be summarized using descriptive statistics by treatment group and total for the ITT population.




A subject data listing of demographics and baseline characteristics will be provided.

#### 4.2 MEDICAL HISTORY

Medical history will be coded with the Medical Dictionary for Regulatory Activities (MedDRA) Terminology version 18.1. The medical history conditions will be summarized by treatment group and total for the safety population using frequencies and percentages on the system organ class (SOC) and preferred term (PT). It also will be presented in the data listings.

# 5. STUDY DRUG AND EXPOSURE

#### 5.1 TREATMENT

A subject data listing will be provided for study drug injection.

#### 5.2 PRIOR AND CONCOMITANT THERAPY

Prior medications are defined as medications that started prior to the intra-articular injection of study drug. Concomitant medications are defined as medications (other than the study drug) taken on or after the intra-articular injection of the study drug during the study. Medications started before the dose of study drug and continuing at the time of the intra-articular injection of study drug are considered both prior medication and concomitant medication.

All investigator terms for medications recorded on the CRF will be coded using the World Health Organization (WHO) Anatomical Therapeutic Chemical (ATC) drug dictionary (Version Dec 2015, WHODDE). The number (percentage) of subjects who took prior and concomitant medications will be summarized in the safety population, by ATC Classification, WHO Drug PT, treatment group and total.

A subject data listing of prior and concomitant therapy will be provided.

# 6. EFFICACY ANALYSES

All efficacy analyses will be performed on the ITT and PP populations.

The primary efficacy hypothesis tests will be performed using a 5% significance level (but, for the MRI improvement evaluation, it shall meet the effective judgment criteria). For the secondary efficacy endpoints, hypothesis tests will be performed individually at the 5% significance level. All hypothesis tests except for the primary efficacy hypothesis tests will be performed with two-sided alternative hypotheses.




# 6.1 PRIMARY EFFICACY ANALYSIS

For primary efficacy endpoints, the joint functional improvement of knee joint will be evaluated using the following three co-primary efficacy variables and gatekeeping procedures will be used for these three hypothesis tests.

Three hypothesis tests will be performed in the following order: 1) Change of WOMAC score within study group, 2) Change of VAS score within study group and 3) MRI improvement evaluation. If null hypothesis is dismissed at 5% significance level for the first hypothesis test, the second hypothesis will also be tested at 5% significance level. Then, for MRI improvement evaluation, the test will be performed to confirm if the percentage of subjects whose final PI evaluation is 'improvement' meets the effective judgment criteria. If null hypothesis is not dismissed at 5% significance level or it is lower than the effective judgment criteria, the hypothesis test is stopped and it is concluded only previous item of which null hypothesis is dismissed is significant.

# 1) Change of WOMAC score from baseline at Month 6 (JointStem group)

Change of WOMAC score from baseline at Month 6 will be tested using paired t-test (one-sided test,  $\alpha$ =0.05) with the null hypothesis equal to zero. The change is defined as WOMAC score at Month 6 minus WOMAC score at baseline. The number of patients, mean, standard deviation, minimum (min) and maximum (max) values for the observed values and change from baseline will be calculated and reported in summary table. In addition, p-value will also be provided. Shapiro-Wilks test will be used to test the normality of change of WOMAC score from baseline at Month 6. If change of WOMAC score from baseline at Month 6 doesn't satisfy normal distribution, Wilcoxon signed rank test will be performed.

If null hypothesis is dismissed, the conclusion that the function of knee joint is improved from at least subjects who administer IP can be drawn.

## 2) Change of VAS score from baseline at Month 6 (JointStem group)

Change of VAS score from baseline at Month 6 will be tested using paired t-test (one-sided test,  $\alpha$ =0.05) with the null hypothesis equal to zero. The change is defined as VAS score at Month 6 minus VAS score at baseline. The number of patients, mean, standard deviation, minimum (min) and maximum (max) values for the observed values and change from baseline will be calculated and reported in summary table. In addition, p-




value will also be provided. Shapiro-Wilks test will be used to test the normality of change of VAS score from baseline at Month 6. If change of VAS score from baseline at Month 6 doesn't satisfy normal distribution, Wilcoxon signed rank test will be performed.

If null hypothesis is dismissed, the conclusion that the pain of degenerative arthritis is reduced from at least subjects who administer IP can be drawn.

# 3) MRI improvement evaluation at Month 6 (JointStem group)

MRI improvement evaluation will be finally analyzed through the following two steps:

- Radiologist will compare and analyze MRI results before and after the administration of IP and write a report for each subject.
- Principal Investigator will evaluate MRI results of subjects as one of three conditions (a: improvement, b: no change, c: progress) based on the radiologist's report stated above.
- → The frequency and percentage of subjects whose final PI evaluation is 'improvement' will be calculated per group.

If the percentage of subjects whose final PI evaluation is at least 36%, the conclusion that the damaged cartilage of knee joint is improved in the subjects who administer JointStem can be drawn.

# 6.2 SECONDARY EFFICACY ANALYSIS

#### 6.2.1 WOMAC Score

WOMAC score will be collected at Visits 3, 4, 5, 6, 7 and 8 (Baseline, M1, M3, M6, M9 and M12) or Early Termination (only if the subject is early terminated after Visit 3) or Final Follow-up Visit. Summary statistics of WOMAC score will be presented by visit and treatment group. The change from baseline will also be calculated and represented in summary table.

- ① Change of WOMAC score from baseline at Month 6 (JointStem group vs. positive control group)
  - This secondary efficacy endpoint will be analyzed with an ANCOVA with factors of treatment and the baseline of WOMAC score as a covariate. Model-based LS Means of the differences between study and control groups, along with 95% CI and p-value will be provided.
- ② Change of WOMAC score from baseline at Months 9 and 12 (JointStem group)




Change of WOMAC score from baseline at Months 9 and 12 will be analyzed using paired t-test (two-sided test,  $\alpha$ =0.05) with the null hypothesis equal to zero. The number of patients, mean, standard deviation, minimum (min) and maximum (max) values for the baseline, months 9, months 12 and change from baseline will be calculated and reported in summary table. The p-value will also be provided. Shapiro-Wilks test will be used to test the normality of change of WOMAC score from baseline at Months 9 and 12. If change of WOMAC score from baseline at Months 9 and 12 doesn't satisfy normal distribution, Wilcoxon signed rank test will be performed.

#### 6.2.2 VAS Score

VAS score will be collected at Visits 3, 4, 5, 6, 7 and 8 (Baseline, M1, M3, M6, M9 and M12) or Early Termination (only if the subject is early terminated after Visit 3) or Final Follow-up Visit. Summary statistics of VAS score will be presented by visit and treatment group. The change from baseline will also be calculated and represented in summary table.

① Change of VAS score from baseline at Month 6 (JointStem group vs. positive control group)

This secondary efficacy endpoint will be analyzed with an ANCOVA with factors of treatment and the baseline of VAS score as a covariate. Model-based LS Means of the differences between study and control groups, along with 95% CI and p-value will be provided.

② Change of VAS score from baseline at Months 9 and 12 (JointStem group)
Change of VAS score from baseline at Months 9 and 12 will be analyzed using paired ttest (two-sided test, α=0.05) with the null hypothesis equal to zero. The number of
patients, mean, standard deviation, minimum (min) and maximum (max) values for the
baseline, months 9, months 12 and change from baseline will be calculated and reported
in summary table. The p-value will also be provided. Shapiro-Wilks test will be used to
test the normality of change of VAS score from baseline at Months 9 and 12. If change
of VAS score from baseline at Months 9 and 12 doesn't satisfy normal distribution,
Wilcoxon signed rank test will be performed.

#### 6.2.3 MRI

① Comparison of MRI improvement evaluations between at Month 6 and at Months 9 and 12 (JointStem group)

MRI improvement evaluation at Month 12 compared to Month 6 will be analyzed using Bowker's test. The frequency and percentage of subjects whose final PI evaluation is




'Improvement' "No change" or "progress" will be calculated at Month 6 and Months 12. The p-value of Bowker's test will be provided.

# 6.2.4 Lysholm Knee Scoring Scale

Lysholm knee scoring scale will be collected at Visits 3, 4, 5, 6, 7 and 8 (Baseline, M1, M3, M6, M9 and M12) or Early Termination (only if the subject is early terminated after Visit 3) or Final Follow-up Visit. Summary statistics of lysholm knee scoring scale will be presented by visit and treatment group. The change from baseline will also be calculated and represented in summary table.

- ① Change of Lysholm Knee Scoring Scale from baseline at Month 6 (JointStem group vs. positive control group)
  - This secondary efficacy endpoint will be analyzed with an ANCOVA with factors of treatment and the baseline of Lysholm Knee Scoring Scale as a covariate. Model-based LS Means of the differences between study and control groups, along with 95% CI and p-value will be provided.
- ② Change of Lysholm Knee Scoring Scale from baseline at Months 6, 9 and 12 (JointStem group)

Change of Lysholm Knee Scoring Scale from baseline at Months 6, 9 and 12 will be analyzed using paired t-test. (two-sided test,  $\alpha$ =0.05) with the null hypothesis equal to zero. The number of patients, mean, standard deviation, minimum (min) and maximum (max) values for the baseline, months 6, months 9, months 12 and change from baseline will be calculated and reported in summary table. The p-value will also be provided. Shapiro-Wilks test will be used to test the normality of change of Lysholm Knee Scoring Scale from baseline at Months 6, 9 and 12. If change of Lysholm Knee Scoring Scale from baseline at Months 6, 9 and 12 doesn't satisfy normal distribution, Wilcoxon signed rank test will be performed.

#### 6.2.5 KOOS

KOOS (Symptoms, Pain, ADL, Sport/Rec, QOL) will be collected at Visits 3, 4, 5, 6, 7 and 8 (Baseline, M1, M3, M6, M9 and M12) or Early Termination (only if the subject is early terminated after Visit 3) or Final Follow-up Visit. Summary statistics of KOOS will be presented by visit and treatment group. The change from baseline will also be calculated and represented in summary table.

① Change of KOOS from baseline at Month 6 (JointStem group vs. positive control group)
This secondary efficacy endpoint will be analyzed with an ANCOVA with factors of




treatment and the baseline of KOOS as a covariate. Model-based LS Means of the differences between study and control groups, along with 95% CI and p-value will be provided.

② Change of KOOS from baseline at Months 6, 9 and 12 (JointStem group)
Change of KOOS from baseline at Months 6, 9 and 12 will be analyzed using paired ttest (two-sided test, α=0.05) with the null hypothesis equal to zero. The number of
patients, mean, standard deviation, minimum (min) and maximum (max) values for the
baseline, months 6, months 9, months 12 and change from baseline will be calculated and
reported in summary table. The p-value will also be provided. Shapiro-Wilks test will be
used to test the normality of change of KOOS from baseline at Months 6, 9 and 12. If
change of KOOS from baseline at Months 6, 9 and 12 doesn't satisfy normal distribution,
Wilcoxon signed rank test will be performed.

#### 6.2.6 IKDC

IKDC will be collected at Visits 3, 4, 5, 6, 7 and 8 (Baseline, M1, M3, M6, M9 and M12) or Early Termination (only if the subject is early terminated after Visit 3) or Final Follow-up Visit. Summary statistics of IKDC will be presented by visit and treatment group. The change from baseline will also be calculated and represented in summary table.

- ① Change of IKDC from baseline at Month 6 (JointStem group vs. positive control group)

  This secondary efficacy endpoint will be analyzed with an ANCOVA with factors of treatment and the baseline of IKDC as a covariate. Model-based LS Means of the differences between study and control groups, along with 95% CI and p-value will be provided.
- ② Change of IKDC from baseline at Months 6, 9 and 12 (JointStem group)
  Change of IKDC from baseline at Months 6, 9 and 12 will be analyzed using paired t-test (two-sided test, α=0.05) with the null hypothesis equal to zero. The number of patients, mean, standard deviation, minimum (min) and maximum (max) values for the baseline, months 6, months 9, months 12 and change from baseline will be calculated and reported in summary table. The 95% CI and p-value will also be provided. Shapiro-Wilks test will be used to test the normality of change of IKDC from baseline at Months 6, 9 and 12. If change of IKDC from baseline at Months 6, 9 and 12 doesn't satisfy normal distribution, Wilcoxon signed rank test will be performed.

#### 6.2.7 RAND-36 Score




RAND-36 Score (Physical Functioning, Role Limitation (Physical), Role Limitation (Emotional), energy/Fatigue, Emotional well-being, Social Functioning, Pain, General Health) at Visits 3, 5, 6, 7 and 8 (Baseline, M3, M6, M9 and M12) or Early Termination (only if the subject is early terminated after Visit 3) or Final Follow-up Visit. Summary statistics of RAND-36 Score will be presented by visit and treatment group. The change from baseline will also be calculated and represented in summary table.

- ① Change of RAND-36 Score from baseline at Month 6 (JointStem group vs. positive control group)
  - This secondary efficacy endpoint will be analyzed with an ANCOVA with factors of treatment and the baseline of RAND-36 Score as a covariate. Model-based LS Means of the differences between study and control groups, along with 95% CI and p-value will be provided.
- ② Change of RAND-36 Score from baseline at Months 6, 9 and 12 (JointStem group) Change of RAND-36 Score from baseline at Months 6, 9 and 12 will be analyzed using paired t-test (two-sided test, α=0.05) with the null hypothesis equal to zero. The number of patients, mean, standard deviation, minimum (min) and maximum (max) values for the baseline, months 6, months 9, months 12 and change from baseline will be calculated and reported in summary table. The 95% CI and p-value will also be provided. Shapiro-Wilks test will be used to test the normality of change of RAND-36 Score from baseline at Months 6, 9 and 12. If change of RAND-36 Score from baseline at Months 6, 9 and 12 doesn't satisfy normal distribution, Wilcoxon signed rank test will be performed.

#### 7. SAFETY ANALYSIS

All safety analyses will be performed for safety population. Statistical tests are not planned for safety variables. Safety assessments include:

- AEs
- Clinical laboratory tests
- ECG
- Physical examinations
- Vital signs

#### 7.1 ADVERSE EVENTS

AEs will be coded by SOC and PT using the MedDRA (Version 18.1). The verbatim term will be included in the AE listing.




A treatment-emergent adverse event (TEAE) is defined as an AE that occur or worsen on or after the injection of study drug and before the end of the study. Only TEAEs will be included in summary tables. All AEs, treatment emergent or otherwise, will be presented in subject data listings.

The TEAEs will be summarized as the number (percentage) of subjects with TEAEs within SOC and PT. Subjects who report the same PT on multiple occasions will be counted once for the PT: under the highest severity (severe > moderate > mild) when summarized by severity and under the closest relationship to study drug when summarized by relationship. If a subject reports multiple PT for a SOC, the subject will be counted only once for that SOC.

TEAEs will be summarized as below.

- An overview table, including number of subjects with
  - o TEAEs
  - o serious AEs (SAEs)
  - o study drug related TEAEs
  - o TEAEs by severity
  - o TEAEs leading to study discontinuation
  - o TEAEs leading to death
- TEAE by SOC and PT
- TEAE by SOC, PT, and Severity
- Study drug related TEAEs by SOC, PT
- SAEs by SOC and PT
- TEAEs leading to study discontinuation by SOC and PT

All AE tables will be sorted by SOC and PT in decreasing frequency of the number and percentage of subjects summarized by treatment group and total.

Missing date will be imputed followed table describes how missing date information will be handled:

| Partial Missing Start or Stop Date | Imputed Start Date | Imputed Stop Date |
|---|---|---|
| Missing month and day, | January 1 of that year or first dose date if the | December 31 of that |
| and the year is present | year is the same as the year of first dose date | year |
| Missing day, but year | First day of that month or first dose date if the | Last day of that |
| and month are present | year and month are the same as the year and | month |
| | month of first dose date | |
| Missing month, but year | Missing month imputed as January | Missing month |
| and day are present | | imputed as December |

# 7.1.1 Deaths, Serious and Other Significant Adverse Events




The listings of serious AEs, AE leading to study discontinuation, and subjects who died during the study will be provided.

#### 7.2 CLINICAL LABORATORY PARAMETERS

Laboratory assessments (hematology, blood chemistry and urinalysis) are collected at Visits 1, 3, 4, 5, 6, 7 and 8 (Screening, Baseline, M1, M3, M6, M9 and M12) or Early Termination (only if the subject is early terminated after Visit 3) or Final Follow-up Visit:

- Chemistry: Total Bilirubin, Alkaline Phosphatase, Aspartate Aminotransferase (AST) (SGPT), Alanine Aminotransferase (ALT) (SGOT), Blood Urea Nitrogen (BUN), Creatinine, Glucose, Albumin, Total protein, Sodium, Potassium, Chloride, Bicarbonate, Calcium, HCG, HIV.
- Hematology: Hemoglobin, Hematocrit, RBC, WBC, MCV, MCH, MCHC, Neutrophils (absolute), Lymphocytes (absolute), Monocytes (absolute), Eosinophils (absolute), Basophils (absolute), Platelets, PT-INR.
- Urinalysis: Specific gravity, Color, Appearance, pH, Protein, Glucose, Ketones, Bilirubin, Blood, Leukocyte esterase, WBC, RBC, Epithelial cell, Bacteria, Hyaline casts.

All laboratory parameters will be presented in Système International (SI) units. Quantitative results (including actual value and change from baseline) will be summarized using descriptive statistics by baseline and post-baseline visit for each laboratory test group above. Laboratory test results were evaluated as normal, abnormal (not clinically significant) or abnormal (clinically significant). The number and percentage of subjects of each category will be summarized by time point, treatment and total for each parameter.

All laboratory data will be included in the listings. A pregnancy listing will be provided separately.

# 7.3 VITAL SIGNS, PHYSICAL EXAMINATIONS FINDINGS, ECG

#### 7.3.1 Vital Signs

Vital signs include sitting blood pressure (BP), pulse, temperature, breathing rate and weight. All vital signs will be presented in Système International (SI) units. Quantitative results (including actual value and change from baseline to each post-baseline visit) will be summarized using descriptive statistics by time point, treatment and total for each parameter.

Listings of vital signs with abnormal flags will be provided.

# 7.3.2 Physical Examinations




Physical examination data will be summarized separately using descriptive statistics by time point, treatment and total, for each component. Listings for physical will be provided.

#### 7.3.3 ECG

The 12-lead ECG parameters including value and changes from baseline will be summarized using descriptive statistics by time point, treatment and total.

Subject listing will be provided. SI units will be used for both summarization and data listings. The critically significant abnormalities will also be flagged in data listings.

# 8. INTERIM ANALYSES AND DATA AND SAFETY MONITORING BOARD (DSMB)

#### 8.1 INTERIM ANALYSES

When at least 15 subjects complete 6-month visits (Visit 6, Month 6), one unblinded interim analysis can be performed to evaluate the efficacy and safety of JointStem without the suspension of subject enrollment. No adjustment on the overall alpha-level will be made, as this is not a statistically powered study. The interim analysis is not covered by this SAP.

#### 8.2 DSMB

No DSMB is planned.

# 9. SUMMARY OF MAJOR CHANGES IN THE PLANNED ANALYSES

There is no major change in the planned analyses based on the study protocol (Version 6.0, Apr 7, 2017).




# **DOCUMENT REVISON HISTORY**

| DATE | VERSION | AUTHOR/ UPDATED BY | COMMENTS |
|----------------|---------|--------------------|---------------------------|
| March 15, 2017 | 1.0 | Hugh Lee | Initial version finalized |
| April 5, 2018 | 2.0 | Byung-Ho Nam | Updated per protocol v6.0 |
